CLINICAL TRIAL: NCT01054534
Title: Real-time Ultrasound Guided Placement of Sacral Quadripolar Leads With Ultrasound Image Fusion of Acquired Magnetic Resonance Scan (MRI)
Brief Title: Ultrasound Image Fusion for Placement of Sacral Quadripolar Leads
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry); Traxtal (Unknown)
Responsible Party: Principal Investigator, Steven R. Clendenen, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-000293
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placement of interstim lead (Other): Placement of interstim lead using US image fusion technology
  Interventions: Procedure: Placement of interstim lead

INTERVENTIONS:
Procedure: Placement of interstim lead — Placement of insterstim lead using US image fusion technology

SUMMARY:
Determine the ability of real-time ultrasound with fusion technology of prior acquired MRI of the pelvis to guide a needle to the second sacral foramen using the posterior approach and place a interstim lead.

ELIGIBILITY:
Inclusion Criteria:

* Patient consented for Interstim lead placement

Exclusion Criteria:

* Patients requesting not to be in the study.
* Pregnant patients

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Identify the third sacral foramen of the pelvis through US image fusion technology | at time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clendenen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States